CLINICAL TRIAL: NCT03833258
Title: A Randomised Controlled Trial of the Impact on Function of an Unrestricted Rehabilitation Pathway of no Precautions Following Total Hip Replacement
Brief Title: Unrestricted Rehabilitation Pathway Following Total Hip Replacement
Acronym: ReHip2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID 19 resulted in cancellation of all elective surgery therefore we need to terminate the trial with 95 participants.
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Justine Theaker, Principal Investigator, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHS001514
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Total Hip Replacement
Keywords: THR; THA; Total Hip Arthroplasty; Total Hip Replacement
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation with precautions (No Intervention): Patients in this arm will continue with rehabilitation following routine care recommendations after total hip replacement; therefore following precautions.
- Rehabilitation with no precautions (Experimental): Patients in this arm will continue with rehabilitation after total hip replacement without precautions, being permitted to move within limits of their own pain only.
  Interventions: Behavioral: Rehabilitation with no precautions

INTERVENTIONS:
Behavioral: Rehabilitation with no precautions — Patients will recover from total hip replacement surgery being guided by pain only and not by the precautions imposed upon them by clinicians.
  Arms: Rehabilitation with no precautions

SUMMARY:
The purpose of ReHip2 is to explore the impact on function and quality of life in patients following Total Hip Replacement (THR). A randomised controlled trial will compare two different rehabilitation pathways following surgery (Routine care with precautions and Treatment group with no precautions). The proposal is to carry out the RCT with a minimum of 182 patients based in the UK.

DETAILED DESCRIPTION:
Dislocation of the hip following total hip replacement (THR) is the sole reason for the endorsement of precautions following THR. This has remained unchanged sine the first hip replacement in 1969.

The precautions are;

* Patients must not bend past 90 degrees at the hip (including sitting)
* Patients must not twist in either standing or sitting
* Patients must partial weight bear with elbow crutches for a minimum of 6 weeks
* Patients must sleep on their back for a minimum of 6 weeks
* Patients must not cross their legs

Studies exploring factors affecting dislocation following THR identified three main influences: surgical technique, type of prosthesis and post-operative precautions. A number of studies have challenged the continued use of precautions or explored their impact on dislocation. However, these studies did not fully consider the impact of all precautions on dislocation, choosing to only select elements of the precautions for investigation. A recent review concluded the evidence evaluating practice and the impact of precautions was of poor quality. The review suggested further research should take into account different surgical approaches, different femoral head sizes and the type of prosthesis. Although there are studies that explored some of these hip dislocation confounders, the true impact of precautions remains unknown.

Whilst precautions continue to be endorsed by surgeons and other clinicians, previous challenges have raised awareness of the possible excessiveness of precautions and the importance of further robust work recommended. This is particularly so in the wake of developments in surgical technique and prostheses design, such as hip joint capsule repair and larger femoral head sizes (larger hip replacements). These developments and their impact on dislocation are beginning to cast doubt on the impact of post-operative precautions and their direct link to incidence of dislocation, which is their primary purpose.

The imposition of precautions has been evidenced to impact on both function and quality of life, with resultant non adherence in a proportion of patients. This study intends to explore whether an unrestricted pathway has no worse outcome in function, pain and quality of life parameters, in two specialist units in a multi-centre, prospective, randomised, non-inferiority study.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants over the age of 18 years will be included.
* All participants should be proceeding with routine care unilateral (one side only) primary THR for treatment of osteoarthritis
* The patients operating consultant agreed to involvement of their patients in the study.
* All subjects assessed during routine pre-operative assessment in their respective hospital will have been assigned an American Society of Anesthesiologists (ASA) up to grade 3 out of a total of 6 (defined as 'severe systemic disease that limits activity but is not incapacitating').
* Patients who have undergone previous hip injection for treatment of osteoarthritic symptoms.
* All surgical approaches (anterior, lateral and posterior), cemented and un-cemented prostheses and all size femoral head size.

Exclusion Criteria:

* The operating consultant declined participation in the study.
* The participant previously had hip surgery to the same hip, including arthroscopy, revision hip surgery or treatment for Avascular Necrosis.
* ASA grade 4 or above 'A patient with severe systemic disease that is a constant threat to life.'
* Patients with specifically identified increased risk of dislocation (for example neuromuscular disease, hypermobility)
* Complex primary hip replacement (THR with femoral osteotomy or structural bone grafting / augmentation of acetabulum)
* Patients unable to complete the postal outcome measures.
* Any patient with pre-operative cognitive impairment (Dementia or Learning disabilities).
* Patients undergoing THR for treatment of fractured neck of femur.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Oxford Hip Score (OHS) | assessed at baseline, 6 and 12 weeks after total hip replacement to assess change at each time point following surgery
  Consists of 12 items measuring pain, activity, joint mobility and ambulatory activity using a 5 point ordinal Likert Scale over the previous 4 weeks. The total score for the OHS range from 12-60 with the lowest score of 12 signifying the least limited function and the highest score of 60 signifying the most limited function.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | assessed at baseline 6 and 12 weeks after total hip replacement to assess change at each time point following surgery
  The Pittsburgh Sleep Quality Index (PSQI) is an outcome measure designed to assess sleep quality, disturbance and impact on function over the preceding one month. The PSQI measures seven categories. Scores total greater than 5 indicate clinically meaningfully disturbed sleep or poor sleep, less than 4 indicates no problems with sleep
EQ-5D-L | assessed at baseline 6 and 12 weeks after total hip replacement to assess change at each time point following surgery
  The lowest score of 0 indicates no functional impairment and a score of 4 indicates significant impairment. The category responses are not combined.
  Using a continuous scale on a 20cm vertical visual analogue scale (VAS) a score of 100 means 'the best health imaginable and a score of 0 means 'the worst health imaginable.' EQ5DL Scores at different timepoints are compared to show changes in health over time

CONTACTS AND LOCATIONS:
Overall Officials: JACQUELINE OLDHAM, Study Chair — University of Manchester
Locations (2):
- United Kingdom (2):
  - Manchester University NHS Foundation Trust, Manchester
  - Wrightington Wigan and Leigh NHS Foundation Trust, Wigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blom AW, Rogers M, Taylor AH, Pattison G, Whitehouse S, Bannister GC. Dislocation following total hip replacement: the Avon Orthopaedic Centre experience. Ann R Coll Surg Engl. 2008 Nov;90(8):658-62. doi: 10.1308/003588408X318156. Epub 2008 Sep 30. PMID 18828962
- [Background] Berry DJ, von Knoch M, Schleck CD, Harmsen WS. Effect of femoral head diameter and operative approach on risk of dislocation after primary total hip arthroplasty. J Bone Joint Surg Am. 2005 Nov;87(11):2456-63. doi: 10.2106/JBJS.D.02860. PMID 16264121
- [Background] Berry DJ, von Knoch M, Schleck CD, Harmsen WS. The cumulative long-term risk of dislocation after primary Charnley total hip arthroplasty. J Bone Joint Surg Am. 2004 Jan;86(1):9-14. doi: 10.2106/00004623-200401000-00003. PMID 14711939
- [Background] Charnley J. Total hip replacement by low-friction arthroplasty. Clin Orthop Relat Res. 1970 Sep-Oct;72:7-21. No abstract available. PMID 5459811
- [Background] Smith TO, Jepson P, Beswick A, Sands G, Drummond A, Davis ET, Sackley CM. Assistive devices, hip precautions, environmental modifications and training to prevent dislocation and improve function after hip arthroplasty. Cochrane Database Syst Rev. 2016 Jul 4;7(7):CD010815. doi: 10.1002/14651858.CD010815.pub2. PMID 27374001
- [Background] Ververeli PA, Lebby EB, Tyler C, Fouad C. Evaluation of reducing postoperative hip precautions in total hip replacement: a randomized prospective study. Orthopedics. 2009 Dec;32(12):889. doi: 10.3928/01477447-20091020-09. PMID 19968217
- [Background] Restrepo C, Mortazavi SM, Brothers J, Parvizi J, Rothman RH. Hip dislocation: are hip precautions necessary in anterior approaches? Clin Orthop Relat Res. 2011 Feb;469(2):417-22. doi: 10.1007/s11999-010-1668-y. PMID 21076896
- [Background] Soong M, Rubash HE, Macaulay W. Dislocation after total hip arthroplasty. J Am Acad Orthop Surg. 2004 Sep-Oct;12(5):314-21. doi: 10.5435/00124635-200409000-00006. PMID 15469226
- [Background] Sharma V, Morgan PM, Cheng EY. Factors influencing early rehabilitation after THA: a systematic review. Clin Orthop Relat Res. 2009 Jun;467(6):1400-11. doi: 10.1007/s11999-009-0750-9. Epub 2009 Mar 10. PMID 19277807
- [Background] Mikkelsen LR, Petersen MK, Soballe K, Mikkelsen S, Mechlenburg I. Does reduced movement restrictions and use of assistive devices affect rehabilitation outcome after total hip replacement? A non-randomized, controlled study. Eur J Phys Rehabil Med. 2014 Aug;50(4):383-93. Epub 2014 Jan 30. PMID 24476806
- [Background] Duwelius PJ, Burkhart RL, Hayhurst JO, Moller H, Butler JB. Comparison of the 2-incision and mini-incision posterior total hip arthroplasty technique: a retrospective match-pair controlled study. J Arthroplasty. 2007 Jan;22(1):48-56. doi: 10.1016/j.arth.2006.09.012. PMID 17197308
- [Background] Jolles BM, Bogoch ER. Posterior versus lateral surgical approach for total hip arthroplasty in adults with osteoarthritis. Cochrane Database Syst Rev. 2004;(1):CD003828. doi: 10.1002/14651858.CD003828.pub2. PMID 14974039
- [Background] Krotenberg R, Stitik T, Johnston MV. Incidence of dislocation following hip arthroplasty for patients in the rehabilitation setting. Am J Phys Med Rehabil. 1995 Nov-Dec;74(6):444-7. doi: 10.1097/00002060-199511000-00010. PMID 8534389
- [Background] Masaoka T, Yamamoto K, Shishido T, Katori Y, Mizoue T, Shirasu H, Nunoda D. Study of hip joint dislocation after total hip arthroplasty. Int Orthop. 2006 Feb;30(1):26-30. doi: 10.1007/s00264-005-0032-4. Epub 2005 Dec 13. PMID 16344996
- [Background] Barnsley L, Barnsley L, Page R. Are Hip Precautions Necessary Post Total Hip Arthroplasty? A Systematic Review. Geriatr Orthop Surg Rehabil. 2015 Sep;6(3):230-5. doi: 10.1177/2151458515584640. PMID 26328242
- [Background] Schmidt-Braekling T, Waldstein W, Akalin E, Benavente P, Frykberg B, Boettner F. Minimal invasive posterior total hip arthroplasty: are 6 weeks of hip precautions really necessary? Arch Orthop Trauma Surg. 2015 Feb;135(2):271-274. doi: 10.1007/s00402-014-2146-x. Epub 2015 Jan 4. PMID 25556661
- [Background] Peak EL, Parvizi J, Ciminiello M, Purtill JJ, Sharkey PF, Hozack WJ, Rothman RH. The role of patient restrictions in reducing the prevalence of early dislocation following total hip arthroplasty. A randomized, prospective study. J Bone Joint Surg Am. 2005 Feb;87(2):247-53. doi: 10.2106/JBJS.C.01513. PMID 15687143
- [Background] Talbot NJ, Brown JH, Treble NJ. Early dislocation after total hip arthroplasty: are postoperative restrictions necessary? J Arthroplasty. 2002 Dec;17(8):1006-8. doi: 10.1054/arth.2002.34534. PMID 12478510
- [Background] Gromov K, Troelsen A, Otte KS, Orsnes T, Ladelund S, Husted H. Removal of restrictions following primary THA with posterolateral approach does not increase the risk of early dislocation--reply. Acta Orthop. 2015;86(4):518-9. No abstract available. PMID 26413601
- [Background] Brooks PJ. Dislocation following total hip replacement: causes and cures. Bone Joint J. 2013 Nov;95-B(11 Suppl A):67-9. doi: 10.1302/0301-620X.95B11.32645. PMID 24187356
- [Background] Jorgensen CC, Kjaersgaard-Andersen P, Solgaard S, Kehlet H; Lundbeck Foundation Centre for Fast-track Hip and Knee Replacement Collaborative Group. Hip dislocations after 2,734 elective unilateral fast-track total hip arthroplasties: incidence, circumstances and predisposing factors. Arch Orthop Trauma Surg. 2014 Nov;134(11):1615-22. doi: 10.1007/s00402-014-2051-3. Epub 2014 Aug 14. PMID 25118616
- [Background] Alberton GM, High WA, Morrey BF. Dislocation after revision total hip arthroplasty : an analysis of risk factors and treatment options. J Bone Joint Surg Am. 2002 Oct;84(10):1788-92. PMID 12377909
- [Background] Ahmad MA, Xypnitos FN, Giannoudis PV. Measuring hip outcomes: common scales and checklists. Injury. 2011 Mar;42(3):259-64. doi: 10.1016/j.injury.2010.11.052. Epub 2010 Dec 15. PMID 21163481
- [Background] Ashby E, Grocott MP, Haddad FS. Outcome measures for orthopaedic interventions on the hip. J Bone Joint Surg Br. 2008 May;90(5):545-9. doi: 10.1302/0301-620X.90B5.19746. PMID 18450615
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Buysse DJ, Yu L, Moul DE, Germain A, Stover A, Dodds NE, Johnston KL, Shablesky-Cade MA, Pilkonis PA. Development and validation of patient-reported outcome measures for sleep disturbance and sleep-related impairments. Sleep. 2010 Jun;33(6):781-92. doi: 10.1093/sleep/33.6.781. PMID 20550019
- [Background] Bystrom S, Espehaug B, Furnes O, Havelin LI; Norwegian Arthroplasty Register. Femoral head size is a risk factor for total hip luxation: a study of 42,987 primary hip arthroplasties from the Norwegian Arthroplasty Register. Acta Orthop Scand. 2003 Oct;74(5):514-24. doi: 10.1080/00016470310017893. PMID 14620970
- [Background] Conner-Spady BL, Marshall DA, Bohm E, Dunbar MJ, Noseworthy TW. Comparing the validity and responsiveness of the EQ-5D-5L to the Oxford hip and knee scores and SF-12 in osteoarthritis patients 1 year following total joint replacement. Qual Life Res. 2018 May;27(5):1311-1322. doi: 10.1007/s11136-018-1808-5. Epub 2018 Feb 8. PMID 29423757
- [Background] Cummins JS, Weinstein JN. The role of patient restrictions in reducing the prevalence of early dislocation following total hip arthroplasty. J Bone Joint Surg Am. 2005 Nov;87(11):2587; author reply 2587-8. doi: 10.2106/00004623-200511000-00028. No abstract available. PMID 16264136
- [Background] Etienne A, Cupic Z, Charnley J. Postoperative dislocation after Charnley low-friction arthroplasty. Clin Orthop Relat Res. 1978 May;(132):19-23. PMID 567107
- [Background] Fielden JM, Gander PH, Horne JG, Lewer BM, Green RM, Devane PA. An assessment of sleep disturbance in patients before and after total hip arthroplasty. J Arthroplasty. 2003 Apr;18(3):371-6. doi: 10.1054/arth.2003.50056. PMID 12728433
- [Background] Forster FJ. Relaxing hip precautions increased patient satisfaction and promoted quicker return to normal activities after total hip arthroplasty. Evid Based Nurs. 2005 Oct;8(4):115. doi: 10.1136/ebn.8.4.115. No abstract available. PMID 16247896
- [Background] Gibbons E, Hewitson P, Morley D, Jenkinson C, Fitzpatrick R. The Outcomes and Experiences Questionnaire: development and validation. Patient Relat Outcome Meas. 2015 Jul 16;6:179-89. doi: 10.2147/PROM.S82784. eCollection 2015. PMID 26213480